CLINICAL TRIAL: NCT05694416
Title: Etoposide Plus Cisplatin Compared With Temozolomide in Patients With Newly Diagnosed MGMT Promotor Unmethylated Glioblastoma
Brief Title: Etoposide Plus Cisplatin Compared With Temozolomide in Patients With Glioblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUTURE
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: MGMT-Unmethylated Glioblastoma
Keywords: Etoposide Plus Cisplatin; Temozolomide; MGMT-Unmethylated Glioblastoma
MeSH Terms: interventions — Etoposide; Cisplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etoposide Plus Cisplatin group (Experimental): Etoposide 100mg/m2 d1-5 Cisplatin 20mg/mCisplatin d1-5
  Interventions: Drug: Etoposide Plus Cisplatin
- Temozolomide group (No Intervention): Temozolomide 150-200mg/m2 d1-5

INTERVENTIONS:
Drug: Etoposide Plus Cisplatin — Etoposide Plus Cisplatin ivdrip d1-5
  Other Names: EP
  Arms: Etoposide Plus Cisplatin group

SUMMARY:
Temozolomide provided significant and clinically meaningful benefit in MGMT gene promoter methylation glioblastoma. However, in unmethylated patients, the effect of Temozolomide is limited. The aim of this study is to compare the effect of Etoposide plus Cisplatin and Temozolomide in patients with MGMT gene promoter unmethylation glioblastoma.

DETAILED DESCRIPTION:
60 Patients with glioblastoma were recruited for this study based on the following eligibility criteria: Age between 18 and 70, performance status of 0-1 (Eastern Cooperative Oncology Group performance status), histologically confirmed MGMT gene promoter unmethylation glioblastoma, no cerebrospinal fluid and distant metastatic disease. All patients had adequate hematologic, hepatic, and renal function. Patients younger than 18 years; patients with a prior (i.e. within 5 years) or synchronous malignancy, other than non-melanoma skin cancer; and those with significant comorbidities were excluded.

60 patients were randomly divided into two groups and compared the difference of efficacy between the two groups

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70,
* performance status of 0-1 (Eastern Cooperative Oncology Group performance status),
* histologically confirmed MGMT gene promoter unmethylation glioblastoma
* no cerebrospinal fluid and distant metastatic disease.
* adequate hematologic, hepatic, and renal function

Exclusion Criteria:

* younger than 18 years;
* with a prior (i.e. within 5 years) or synchronous malignancy, other than non-melanoma skin cancer; and those with significant comorbidities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
OVER SURVIVAL | 2 YEARS
  The length of time from the date of diagnosis to death from cancer

SECONDARY OUTCOMES:
PFS | 1 year
  the length of time after primary treatment for glioblastoma ends that the patient survives without any progression of glioblastoma.

CONTACTS AND LOCATIONS:
Overall Officials: Jianyin Huang, MD, Study Chair — Wuhan University